CLINICAL TRIAL: NCT01153347
Title: A Multicenter, Randomized, Double-Blind Parallel Group Placebo-Controlled Phase III,Efficacy and Safety Study of 3 Fixed Dose Groups of TC-5214 (S-mecamylamine) as an Adjunct to an Antidepressant in Patients With Major Depressive Disorder Who Exhibit an Inadequate Response to Antidepressant Therapy
Brief Title: A Study to Assess the Efficacy and Safety of TC-5214 as an Adjunct Therapy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4130C00004
Record Dates: First submitted 2010-06-23; First posted 2010-06-30 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Major Depressive Disorder; Depression
Keywords: Major Depressive Disorder; MDD; Depression; Safety; add-on therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SSRI/Serotonin/SNRI+ TC-5214 0.5 mg (Experimental): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 0.5 mg BID
  Interventions: Drug: TC-5214
- SSRI/Serotonin/SNRI + TC-5214 2 mg (Experimental): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 2 mg BID
  Interventions: Drug: TC-5214
- SSRI/Serotonin/SNRI + TC-5214 4 mg (Experimental): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 4 mg BID
  Interventions: Drug: TC-5214
- SSRI/Serotonin/SNRI + Placebo (Placebo Comparator): Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — Tablet, oral, twice daily for 8 weeks
  Arms: SSRI/Serotonin/SNRI + TC-5214 2 mg; SSRI/Serotonin/SNRI + TC-5214 4 mg; SSRI/Serotonin/SNRI+ TC-5214 0.5 mg
Drug: Placebo — Tablet, oral, twice daily for 8 weeks
  Arms: SSRI/Serotonin/SNRI + Placebo

SUMMARY:
The purpose of this study is to determine if TC-5214 or placebo (a tablet that looks like medicine tablet or capsule, but contains no active medicine) is safe and effective when taken together with another antidepressant.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures.
* The patient must have a clinical diagnosis of major depressive disorder (MDD) with inadequate response to no more than one antidepressant.
* Outpatient status at enrollment and randomization.

Exclusion Criteria:

* Patients with a lifetime history of bipolar disorder, psychotic disorder or post-traumatic stress disorder.
* Patients with a history of suicide attempts in the past year and/or seen by the investigator as having a significant history of risk of suicide or homicide.
* History of renal insufficiency or impairment or conditions that could affect absorption or metabolism of investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2409 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans A. Eriksson, MD,PhD, MBA, Study Director — AstraZeneca; Andrew J. Cutler, MD, Principal Investigator — Florida Clinical Research Center, LLC
Locations (99):
- United States (79):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Conway, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Arcadia, California
  - Research Site, Beverly Hills, California
  - Research Site, Garden Grove, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Oakland, California
  - Research Site, Oceanside, California
  - Research Site, Pico Rivera, California
  - Research Site, Santa Ana, California
  - Research Site, Upland, California
  - Research Site, Denver, Colorado
  - Research Site, Cromwell, Connecticut
  - Research Site, New London, Connecticut
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bradenton, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Fort Walton Beach, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Plantation, Florida
  - Research Site, South Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Valparaiso, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Florence, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Gaithersburg, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Weymouth, Massachusetts
  - Research Site, Flowood, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, North Platte, Nebraska
  - Research Site, Toms River, New Jersey
  - Research Site, Willingboro, New Jersey
  - Research Site, Mount Kisco, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Avon Lake, Ohio
  - Research Site, Beachwood, Ohio
  - Research Site, Beechwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Mason, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sellersvillle, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Murray, Utah
  - Research Site, Bellevue, Washington
  - Research Site, Bothell, Washington
  - Research Site, Seattle, Washington
  - Research Site, South Kirkland, Washington
  - Research Site, Spokane, Washington
- India (19):
  - Research Site, Guntur, Andhra Pradesh
  - Research Site, Vijayawada, Andhra Pradesh
  - Research Site, Visakhapatnam, Andhra Pradesh
  - Research Site, Anand, Gujarat
  - Research Site, Jūnāgadh, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Aurangabad, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Nashik, Mahara
  - Research Site, Durham, NC
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Varanasi, Uttar Prad
  - Research Site, Kanpur
  - Research Site, Karnataka
  - Research Site, Mysore
- Research Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Moller HJ, Demyttenaere K, Olausson B, Szamosi J, Wilson E, Hosford D, Dunbar G, Tummala R, Eriksson H. Two Phase III randomised double-blind studies of fixed-dose TC-5214 (dexmecamylamine) adjunct to ongoing antidepressant therapy in patients with major depressive disorder and an inadequate response to prior antidepressant therapy. World J Biol Psychiatry. 2015 Oct;16(7):483-501. doi: 10.3109/15622975.2014.989261. Epub 2015 Jan 20. PMID 25602163
- See also: CSR-D4130C00004.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=2777&filename=CSR-D4130C00004.pdf
- See also: D4130C00004/Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2777&filename=D4130C00004_Revised_CSP_1_redacted_13Nov13.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in the US and India between 15 June 2010 and 31 January 2012.
Pre-assignment Details: The study had an up to 21-day screening/washout period, and an 8-week prospective open-label antidepressant treatment (ADT) period to identify the target patient population of inadequate responders to ADT (<50% reduction in HAMD-17 total score during the prospective open-label ADT period, a HAMD-17 total score of ≥16 and a CGI-S score ≥4).
Groups:
- 0.5 mg BID TC-5214: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 0.5 mg BID
- 2 mg BID TC-5214: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 2 mg BID
- 4 mg BID TC-5214: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + TC-5214, 4 mg BID
- Placebo: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + Placebo BID
Period: Overall Study
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Started | 160 | 160 | 160 | 161
Received Treatment | 160 | 158 | 158 | 160
Completed | 127 | 116 | 110 | 129
Not Completed | 33 | 44 | 50 | 32
Not completed — Withdrawal by Subject | 7 | 7 | 7 | 7
Not completed — Eligibility criteria not fulfilled | 0 | 1 | 2 | 1
Not completed — Adverse Event | 3 | 9 | 21 | 7
Not completed — Severe non-compliance to protocol | 6 | 7 | 4 | 3
Not completed — Condition under investigation worsened | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 0 | 4
Not completed — Study-specific withdrawal criteria | 4 | 3 | 1 | 2
Not completed — Lost to Follow-up | 4 | 9 | 11 | 8
Not completed — Other | 5 | 5 | 4 | 0
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo | Total
Number analyzed (Participants) | 160 | 160 | 160 | 161 | 641
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (11.78) | 42.1 (11.77) | 42.1 (11.35) | 43.2 (11.92) | 42.0 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 91 | 93 | 96 | 365
  Male | 75 | 69 | 67 | 65 | 276
Race/Ethnicity, Customized [Number; unit: participants]
  White | 87 | 100 | 91 | 103 | 381
  Black or African American | 20 | 23 | 27 | 14 | 84
  Asian | 50 | 35 | 40 | 42 | 167
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Other | 3 | 1 | 2 | 1 | 7
Hamilton Rating Scale for Depression-17 items (HAMD-17) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
  Scores on a scale | 22.3 (3.98) | 21.5 (3.74) | 22.0 (4.07) | 22.1 (4.08) | 22.0 (3.97)
Montgomery-Asberg Depression Rating Scale (MADRS) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
  Scores on a scale | 26.86 (6.331) | 26.37 (6.036) | 27.06 (5.854) | 26.70 (6.809) | 26.75 (6.261)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Randomization to End of Treatment.
Description: A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: Modified intent-to-treat analysis set including all randomized patients who received at least 1 dose of investigational product (TC-5214 or placebo) and who had a randomization and at least 1 post-randomization MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 155 | 156 | 152 | 157
units on a scale | -12.1 (0.81) | -11.8 (0.83) | -11.3 (0.84) | -11.2 (0.80)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; Mixed model repeated measures (MMRM) includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 1.000, MMRM — The adjusted p-value protects the overall family-wise error rate by taking into account the multiple comparisons between the TC-5214 doses for both the primary efficacy variable (MADRS) and the key secondary efficacy variable (SDS); LS mean = -0.9, 95% CI 2-sided [-2.96 to 1.24], Standard Error of Mean 1.07
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM; LS mean = -0.6, 95% CI 2-sided [-2.67 to 1.57], Standard Error of Mean 1.08
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM; LS mean = -0.1, 95% CI 2-sided [-2.26 to 2.04], Standard Error of Mean 1.09

2. Secondary Outcome: Response in Depressive Symptoms of Major Depressive Disorder (MDD), Defined as a ≥50% Reduction From Randomization (Week 8) in MADRS Total Score at End of Treatment (Week 16)
Description: The percentage of patients with a ≥50% reduction from randomization (Week 8) in MADRS total score at end of treatment (Week 16) was calculated.
  A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 155 | 156 | 152 | 157
percentage of participants analyzed | 43.9 | 39.7 | 38.8 | 42.7
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; Logistic regression model including treatment and pooled center as fixed effects and the randomization MADRS total score as a covariate; Test type: Superiority or Other; p = 0.967, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.64 to 1.60], Standard Error of Mean 0.24 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.670, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.57 to 1.43], Standard Error of Mean 0.21 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.544, Regression, Logistic; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.54 to 1.38], Standard Error of Mean 0.21 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

3. Secondary Outcome: Remission in Depressive Symptoms of MDD, Defined as MADRS Total Score of ≤8 at End of Treatment (Week 16)
Description: The percentage of patients with a MADRS total score of ≤8 at end of treatment (Week 16) was calculated.
  A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 155 | 156 | 152 | 157
percentage of participants analyzed | 29.0 | 26.9 | 23.7 | 29.9
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.730, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.55 to 1.53], Standard Error of Mean 0.24 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.671, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.53 to 1.50], Standard Error of Mean 0.23 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.308, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.45 to 1.29], Standard Error of Mean 0.20 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

4. Secondary Outcome: Early and Sustained Response, Defined as a ≥50% Reduction From Randomization (Week 8) in MADRS Total Score and a MADRS Total Score of ≤12 at Week 10, Week 12, Week 14, and End of Treatment (Week 16)
Description: The percentage of patients with a ≥50% reduction from randomization (Week 8) in MADRS total score and a MADRS total score of ≤12 at Week 10, Week 12, Week 14, and end of treatment (Week 16) was calculated.
  A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16); Week 10, Week 12, Week 14, and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 148 | 153 | 145 | 153
percentage of participants analyzed | 8.8 | 7.8 | 8.3 | 8.5
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.905, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.42 to 2.15], Standard Error of Mean 0.40 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.864, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.41 to 2.14], Standard Error of Mean 0.39 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.958, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.43 to 2.25], Standard Error of Mean 0.42 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

5. Secondary Outcome: Sustained Response, Defined as a ≥50% Reduction From Randomization (Week 8) in MADRS Total Score and a MADRS Total Score of ≤12 at Week 12, Week 14, and End of Treatment (Week 16)
Description: The percentage of patients with a ≥50% reduction from randomization (Week 8) in MADRS total score and a MADRS total score of ≤12 at Week 12, Week 14, and end of treatment (Week 16) was calculated.
  A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16); Week 12, Week 14, and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of patients analyzed
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 145 | 150 | 143 | 151
percentage of patients analyzed | 15.9 | 18.7 | 14.0 | 15.9
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.778, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.48 to 1.73], Standard Error of Mean 0.30 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.532, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.66 to 2.24], Standard Error of Mean 0.38 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.633, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.44 to 1.64], Standard Error of Mean 0.29 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

6. Secondary Outcome: Sustained Remission, Defined as a MADRS Total Score of ≤8 at Week 12, Week 14, and End of Treatment (Week 16)
Description: The percentage of patients with a MADRS total score of ≤8 at Week 12, Week 14, and end of treatment (Week 16)was calculated.
  A 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Week 12, Week 14, Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 146 | 150 | 144 | 152
percentage of participants analyzed | 10.3 | 12.7 | 7.6 | 9.2
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.949, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.46 to 2.31], Standard Error of Mean 0.42 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.253, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.72 to 3.40], Standard Error of Mean 0.62 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.763, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.37 to 2.08], Standard Error of Mean 0.39 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

7. Secondary Outcome: Change in Depressive Symptoms From Randomization (Week 8) to End of Treatment (Week 16) as Measured by Hamilton Rating Scale for Depression-17 Items (HAMD-17) Total Score
Description: A 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 147 | 144 | 142 | 150
units on a scale | -10.1 (0.79) | -9.7 (0.79) | -9.5 (0.79) | -9.1 (0.78)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; Analysis of covariance (ANCOVA) with randomization HAMD-17 total score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.207, ANCOVA; LS mean = -1.0, 95% CI 2-sided [-2.51 to 0.55], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.427, ANCOVA; LS mean = -0.6, 95% CI 2-sided [-2.16 to 0.91], Standard Error of Mean 0.78
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.591, ANCOVA; LS mean = -0.4, 95% CI 2-sided [-1.96 to 1.12], Standard Error of Mean 0.78

8. Secondary Outcome: Change in the Clinician-rated Global Outcome of Severity as Measured by the Clinical Global Impression-Severity (CGI-S) Score From Randomization (Week 8) to End of Treatment (Week 16)
Description: A 3-part, clinician-administered scale that rates the improvement or worsening of the patient's illness from randomization (baseline). Each item is scored on a 1 to 7 scale. Higher CGI-S scores indicate greater illness severity.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 155 | 156 | 152 | 157
units on a scale | -1.3 (0.10) | -1.3 (0.11) | -1.2 (0.11) | -1.2 (0.10)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit, and treatment by visit interaction as explanatory variables and the randomization CGI-S total score as a covariate. Treatment, visit, and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.551, MMRM; LS mean = -0.1, 95% CI [-0.34 to 0.18], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.487, MMRM; LS mean = -0.1, 95% CI 2-sided [-0.36 to 0.17], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.780, MMRM; LS mean = 0.0, 95% CI 2-sided [-0.23 to 0.31], Standard Error of Mean 0.14

9. Secondary Outcome: Response in the Clinical Global Impression-Improvement (CGI-I) Defined as CGI-I Rating of "Very Much Improved" or "Much Improved" From Randomization (Week 8) to End of Treatment (Week 16)
Description: A 3-part, clinician-administered scale that rates the improvement or worsening of the patient's illness from randomization (baseline). Each item is scored on a 1 to 7 scale. CGI-I scores >4 indicate worsening, while scores <4 indicate improvement.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 155 | 156 | 152 | 157
percentage of participants analyzed | 48.4 | 49.4 | 37.5 | 47.8
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; Logistic regression model including treatment and pooled center as fixed effects and the randomization Clinical Global Impression Severity (CGI-S) as a covariate; Test type: Superiority or Other; p = 0.908, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.62 to 1.53], Standard Error of Mean 0.23 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.803, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.67 to 1.67], Standard Error of Mean 0.24 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.066, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.41 to 1.03], Standard Error of Mean 0.15 — TC-5214 is the numerator in the OR, OR>1 represents a result in favor of TC-5214

10. Secondary Outcome: Change in Hamilton Anxiety Scale (HAM-A) Total Score From Randomization (Week 8) to End of Treatment (Week 16)
Description: A 14-item clinician-administered scale for the evaluation of anxiety symptoms. Each HAM-A item is rated on a 0 to 4 scale, the total score can range from 0 to 56. Higher HAM-A scores indicate higher levels of anxiety.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 147 | 144 | 142 | 150
units on a scale | -7.07 (0.648) | -6.46 (0.652) | -6.75 (0.655) | -6.24 (0.641)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; An analysis of covariance (ANCOVA) with randomization HAM-A total score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.202, ANCOVA; LS mean = -0.82, 95% CI 2-sided [-2.091 to 0.442], Standard Error of Mean 0.645
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.738, ANCOVA; LS mean = -0.22, 95% CI 2-sided [-1.487 to 1.055], Standard Error of Mean 0.647
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.433, ANCOVA; LS mean = -0.51, 95% CI 2-sided [-1.787 to 0.767], Standard Error of Mean 0.650

11. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 9
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 150 | 146 | 152
units on a scale | -4.0 (0.52) | -5.1 (0.52) | -4.0 (0.52) | -5.0 (0.52)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.097, MMRM; LS mean = 1.0, 95% CI 2-sided [-0.18 to 2.22], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.882, MMRM; LS mean = -0.1, 95% CI 2-sided [-1.29 to 1.11], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.100, MMRM; LS mean = 1.0, 95% CI 2-sided [-0.19 to 2.23], Standard Error of Mean 0.62

12. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 10
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 150 | 146 | 139 | 148
units on a scale | -6.3 (0.60) | -6.9 (0.60) | -7.3 (0.61) | -7.1 (0.60)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.303, MMRM; LS mean = 0.8, 95% CI 2-sided [-0.69 to 2.22], Standard Error of Mean 0.74
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.793, MMRM; LS mean = 0.2, 95% CI 2-sided [-1.26 to 1.65], Standard Error of Mean 0.74
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.762, MMRM; LS mean = -0.2, 95% CI 2-sided [-1.70 to 1.25], Standard Error of Mean 0.75

13. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 12
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 142 | 135 | 128 | 145
units on a scale | -9.4 (0.70) | -9.4 (0.71) | -8.9 (0.73) | -8.5 (0.70)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.339, MMRM; LS mean = -0.9, 95% CI 2-sided [-2.65 to 0.92], Standard Error of Mean 0.91
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.321, MMRM; LS mean = -0.9, 95% CI 2-sided [-2.70 to 0.89], Standard Error of Mean 0.91
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.680, MMRM; LS mean = -0.4, 95% CI 2-sided [-2.20 to 1.43], Standard Error of Mean 0.92

14. Secondary Outcome: Change in MADRS Total Score From Randomization (Week 8) to Week 14
Description: as for outcome 1
Time Frame: Randomization (Week 8) to Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 140 | 127 | 119 | 134
units on a scale | -11.0 (0.74) | -11.3 (0.76) | -10.6 (0.77) | -10.7 (0.74)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.737, MMRM; LS mean = -0.3, 95% CI 2-sided [-2.23 to 1.58], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.547, MMRM; LS mean = -0.6, 95% CI 2-sided [-2.52 to 1.33], Standard Error of Mean 0.98
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.953, MMRM; LS mean = 0.1, 95% CI 2-sided [-1.89 to 2.01], Standard Error of Mean 0.99

15. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by the Sheehan Disability Scale (SDS) Total Score
Description: Sheehan Disability Scale (SDS) is 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The SDS total score is calculated as the sum of the score for the 3 inter-correlated domains (school/work, social life, and family life/home responsibilities) and ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 148 | 149 | 153
units on a scale | -5.53 (0.631) | -5.45 (0.643) | -4.53 (0.651) | -4.93 (0.627)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit, and treatment by visit interaction as explanatory variables and the randomization SDS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 1.000, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean = -0.60, 95% CI 2-sided [-2.069 to 0.864], Standard Error of Mean 0.746
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean = -0.52, 95% CI 2-sided [-2.004 to 0.960], Standard Error of Mean 0.755
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 1.000, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean = 0.40, 95% CI 2-sided [-1.095 to 1.896], Standard Error of Mean 0.761

16. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by SDS Work/School Domain Score
Description: A 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The 3 inter-correlated domains are school/work, social life, and family life/home responsibilities. The numerical rating for the work/school domain score is 0- 10, where 10 is considered to be 'highly impaired'.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 132 | 123 | 134 | 137
units on a scale | -1.7 (0.21) | -1.8 (0.22) | -1.7 (0.21) | -1.7 (0.21)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization SDS work/school domain score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.953, MMRM; LS mean = 0.0, 95% CI 2-sided [-0.56 to 0.59], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.868, MMRM; LS mean = 0.0, 95% CI 2-sided [-0.64 to 0.54], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.792, MMRM; LS mean = 0.1, 95% CI 2-sided [-0.50 to 0.66], Standard Error of Mean 0.30

17. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by SDS Social Life Domain Score
Description: A 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The 3 inter-correlated domains are school/work, social life, and family life/home responsibilities. The numerical rating for the SDS social life domain score is 0- 10, where 10 is considered to be 'highly impaired'.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 148 | 149 | 153
units on a scale | -1.9 (0.22) | -1.9 (0.23) | -1.6 (0.23) | -1.9 (0.22)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization SDS social life domain score. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.915, MMRM; LS mean = 0.0, 95% CI 2-sided [-0.54 to 0.48], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.972, MMRM; LS mean = 0.0, 95% CI 2-sided [-0.51 to 0.53], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.237, MMRM; LS mean = 0.3, 95% CI 2-sided [-0.21 to 0.84], Standard Error of Mean 0.27

18. Secondary Outcome: Change in Functional Impairment From Randomization (Week 8) to End of Treatment (Week 16) as Measured by SDS Family Life/Home Responsibilities Domain Score
Description: A 5-item, self-administered scale that measures the extent a patient is impaired by their disease. Higher scores indicate more severe impairment. The 3 inter-correlated domains are school/work, social life, and family life/home responsibilities. The numerical rating for the SDS family life/home responsibilities domain score is 0- 10, where 10 is considered to be 'highly impaired'.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 148 | 149 | 153
units on a scale | -1.9 (0.22) | -1.8 (0.23) | -1.6 (0.23) | -1.6 (0.22)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization SDS family life/home responsibilities domain score. Treatment, visit and treatment by visit interaction are effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.213, MMRM; LS mean = -0.3, 95% CI 2-sided [-0.87 to 0.19], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.343, MMRM; LS mean = -0.3, 95% CI 2-sided [-0.80 to 0.28], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.971, MMRM; LS mean = 0.0, 95% CI 2-sided [-0.55 to 0.53], Standard Error of Mean 0.28

19. Secondary Outcome: Change in Overall Quality of Life and Satisfaction From Randomization (Week 8) to End of Treatment (Week 16) by Assessing the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) % Maximum Total Score
Description: The Q-LES-Q-SF total score is derived by summing item scores 1 to 14. Higher scores are indicative of greater enjoyment or satisfaction in each domain. The Q-LES-Q-SF % maximum total score is calculated as 100% × (Q-LES-Q-SF total score - 14) / 56, and can range from 0% to 100%.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 148 | 144 | 151
units on a scale | 12.81 (1.470) | 11.42 (1.483) | 8.83 (1.499) | 10.71 (1.467)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; ANCOVA with randomization Q-LES-Q-SF % maximum total score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.215, ANCOVA; LS mean = 2.10, 95% CI 2-sided [-1.224 to 5.431], Standard Error of Mean 1.694
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.673, ANCOVA; LS mean = 0.72, 95% CI 2-sided [-2.624 to 4.062], Standard Error of Mean 1.702
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.275, ANCOVA; LS mean = -1.88, 95% CI 2-sided [-5.248 to 1.494], Standard Error of Mean 1.716

20. Secondary Outcome: Change From Randomization (Week 8) to End of Treatment (Week 16) in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form(Q LES-Q-SF)Item 15
Description: The Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form) measures the patient's satisfaction with medication and overall quality of life. The 15th item queries respondents' satisfaction with the medication they are taking, rated on a 1 to 4 scale, score 0 indicates that no medication was taken. Higher scores are indicative of greater satisfaction.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 142 | 136 | 124 | 138
units on a scale | 0.3 (0.08) | 0.4 (0.08) | 0.2 (0.08) | 0.4 (0.08)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; An analysis of covariance (ANCOVA) with randomization Q-LES-Q-SF item 15 score as covariate, treatment as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.412, ANCOVA; LS mean = -0.1, 95% CI 2-sided [-0.28 to 0.11], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.928, ANCOVA; LS mean = 0.0, 95% CI 2-sided [-0.19 to 0.21], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.033, ANCOVA; LS mean = -0.2, 95% CI 2-sided [-0.42 to -0.02], Standard Error of Mean 0.10

21. Secondary Outcome: Change From Randomization (Week 8) to End of Treatment (Week 16) in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q LES-Q-SF) Item 16
Description: The Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form) measures the patient's satisfaction with medication and overall quality of life. The 16th item is a global rating of overall life satisfaction and contentment, rated on a 1 to 5 scale. Higher scores are indicative of greater satisfaction.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 148 | 144 | 151
units on a scale | 0.6 (0.08) | 0.5 (0.08) | 0.4 (0.08) | 0.5 (0.08)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; An analysis of covariance (ANCOVA) with randomization Q-LES-Q-SF item 16 as a fixed effect and pooled center as a random effect; Test type: Superiority or Other; p = 0.353, ANCOVA; LS mean = 0.1, 95% CI 2-sided [-0.10 to 0.28], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.721, ANCOVA; LS mean = 0.0, 95% CI 2-sided [-0.16 to 0.23], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.666, ANCOVA; LS mean = 0.0, 95% CI 2-sided [-0.24 to 0.15], Standard Error of Mean 0.10

22. Secondary Outcome: Change in EuroQol - 5 Dimensions (EQ-5D) From Randomization (Week 8) to End of Treatment (Week 16)
Description: A self-assessment questionnaire that provides 2 measures of health status. The EQ-5D index score is a weighted linear combination over 5 dimensions of health status. The score for each of the 5 dimensions can range from 1 to 3, and an equation is used to calculate the EQ-5D index score. The EQ-5D index score can range from possible negative values (minimum -0.415) to a maximum of 1.0. The EQ-VAS is a visual analog scale with a range of 0 to 100. For both variables, a higher score indicates a better health state.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 147 | 147 | 153
units on a scale
  EQ-5D index score | 0.114 (0.0169) | 0.107 (0.0173) | 0.106 (0.0176) | 0.120 (0.0168)
  EQ-5D VAS score | 13.4 (1.69) | 12.9 (1.73) | 10.3 (1.76) | 11.5 (1.68)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization EQ-5D total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.747, MMRM — Analysis for change in EQ-5D index score from randomization (Week 8) to end of treatment (Week 16); LS mean = -0.006, 95% CI 2-sided [-0.0459 to 0.0329], Standard Error of Mean 0.0201
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.524, MMRM — Analysis for change in EQ-5D index score from randomization (Week 8) to end of treatment (Week 16); LS mean = -0.013, 95% CI 2-sided [-0.0529 to 0.0270], Standard Error of Mean 0.0203
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.502, MMRM — Analysis for change in EQ-5D index score from randomization (Week 8) to end of treatment (Week 16); LS mean = -0.014, 95% CI 2-sided [-0.0543 to 0.0267], Standard Error of Mean 0.0206
Statistical Analysis 4: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit and treatment by visit interaction as explanatory variables and the randomization EQ-5D VAS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.345, MMRM — Analysis of change in EQ-5D VAS score from randomization (Week 8) to end of treatment (Week 16); LS mean = 1.9, 95% CI 2-sided [-2.10 to 6.00], Standard Error of Mean 2.06
Statistical Analysis 5: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Superiority or Other; p = 0.486, MMRM — Analysis of change in EQ-5D VAS score from randomization (Week 8) to end of treatment (Week 16); LS mean = 1.5, 95% CI 2-sided [-2.65 to 5.56], Standard Error of Mean 2.09
Statistical Analysis 6: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 22, analysis 4]; Test type: Superiority or Other; p = 0.564, MMRM — Analysis of change in EQ-5D VAS score from randomization (Week 8) to end of treatment (Week 16); LS mean = -1.2, 95% CI 2-sided [-5.39 to 2.94], Standard Error of Mean 2.12

23. Secondary Outcome: Change in Irritability Symptoms as Measured by the Sheehan Irritability Scale (SIS) Total Score From Randomization (Week 8) to End of Treatment (Week 16)
Description: A self-administered scale to be used by clinical subjects to rate suffering over the past week with regard to irritability symptoms. The total SIS score is the sum of 7 items, and ranges from 0 to 70. Each item is assessed on an 11- point scale where 0=not at all, 1-3=mildly, 4-6=moderately, 7-9=markedly, and 10=extremely. The SIS also records the number of days impaired by irritability.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214 | Placebo
Number analyzed (Participants) | 152 | 148 | 149 | 153
units on a scale | -10.2 (1.46) | -10.1 (1.49) | -8.3 (1.50) | -8.8 (1.46)
Statistical Analysis 1: Comparison: 0.5 mg BID TC-5214 vs Placebo; MMRM model includes treatment, pooled center, visit, and treatment by visit interaction as explanatory variables and the randomization SIS total score as a covariate. Treatment, visit and treatment by visit interaction are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.350, MMRM; LS mean = -1.4, 95% CI 2-sided [-4.48 to 1.59], Standard Error of Mean 1.55
Statistical Analysis 2: Comparison: 2 mg BID TC-5214 vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.393, MMRM; LS mean = -1.3, 95% CI 2-sided [-4.41 to 1.73], Standard Error of Mean 1.56
Statistical Analysis 3: Comparison: 4 mg BID TC-5214 vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.745, MMRM; LS mean = 0.5, 95% CI 2-sided [-2.59 to 3.62], Standard Error of Mean 1.58

ADVERSE EVENTS:
Groups:
- Placebo: Selective serotonin reuptake inhibitor (SSRI)/Serotonin/norepinephrine reuptake inhibitor (SNRI) + Placebo
Arm/Group | Placebo | 0.5 mg BID TC-5214 | 2 mg BID TC-5214 | 4 mg BID TC-5214
Serious Adverse Events (participants affected / at risk) | 2/160 | 2/160 | 0/158 | 5/158
Other Adverse Events (participants affected / at risk) | 76/160 | 80/160 | 88/158 | 99/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=160) | 0.5 mg BID TC-5214 (N=160) | 2 mg BID TC-5214 (N=158) | 4 mg BID TC-5214 (N=158)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scapula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive Uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=160) | 0.5 mg BID TC-5214 (N=160) | 2 mg BID TC-5214 (N=158) | 4 mg BID TC-5214 (N=158)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (7)
Constipation (Gastrointestinal disorders) | 7 (8) | 12 (13) | 25 (28) | 45 (48)
Nausea (Gastrointestinal disorders) | 10 (11) | 7 (7) | 13 (13) | 10 (11)
Dry Mouth (Gastrointestinal disorders) | 2 (3) | 6 (6) | 11 (11) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 10 (11) | 8 (8) | 10 (11)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 5 (6) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (5) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
Fatigue (General disorders) | 6 (6) | 2 (2) | 4 (4) | 7 (8)
Pyrexia (General disorders) | 1 (2) | 5 (5) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Pain (General disorders) | 3 (3) | 4 (4) | 1 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 7 (7) | 6 (6) | 7 (8) | 5 (5)
Bronchitis (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 2 (2) | 6 (6) | 3 (3)
Sinusitis (Infections and infestations) | 4 (5) | 2 (2) | 3 (3) | 0 (0)
Aspartate Aminotransferase Increased (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 22 (25) | 14 (19) | 15 (17) | 13 (14)
Dizziness (Nervous system disorders) | 3 (3) | 11 (11) | 8 (8) | 14 (14)
Somnolence (Nervous system disorders) | 5 (5) | 6 (6) | 4 (4) | 8 (8)
Dizziness Postural (Nervous system disorders) | 2 (2) | 1 (1) | 3 (5) | 5 (7)
Akathisia (Nervous system disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (10) | 8 (8) | 8 (8) | 6 (7)
Abnormal Dreams (Psychiatric disorders) | 3 (3) | 2 (2) | 6 (6) | 2 (2)
Agitation (Psychiatric disorders) | 4 (4) | 5 (5) | 4 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Orthostatic Hypotension (Vascular disorders) | 2 (3) | 1 (1) | 1 (5) | 5 (5)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days